CLINICAL TRIAL: NCT04040556
Title: Enhancing Student Learning by Simulation
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Primary investigator, Prince of Songkla University
Other Study IDs: Simulation SDL
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Pre and Post Simulation Session Self-directed Learning Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesia residence: anesthesia residences who currently study in the department of Anesthesia and voluntarily enrolled into the study
  Interventions: Other: Simulation class

INTERVENTIONS:
Other: Simulation class — Pediatric anesthesia simulation class for anesthesia residences
  Other Names: Simulation session

SUMMARY:
As the standard of best practice, care of complicated or difficult patient needs not only knowledge but also including skills and clinical thinking in many aspects.

Simulation is now accepted as the way of teaching for adult learners. This learning method can help students to apply their knowledge, practical skills and non-technical skills. A systematic review study showed that self-directed learning (SDL) in health professions education is associated with moderate improvement in the knowledge domain. SDL also help the learners to improve self-efficacy and the learning outcomes in complicated tasks.In this study, the investigators wanted to evaluate that simulation can enhance student to do SDL in the both pre and post session period.

DETAILED DESCRIPTION:
After approval from the instution's Ethics Committee, a prospective cohort study was conducted between November 2017 to March 2018. Twenty-five anesthesia residents were participated in this study. Students were noticed about the simulation classes which are emergencies in pediatric anesthesia and complications at one-month prior the day of practice. The list of standard references was given. On the day of study, at the institute's simulation center, students were voluntarily separated into two groups, directed- learner and observer. Post class debriefing sessions were done as routine activities. After the class, the investigator invited the students to be enrolled in this study by using the flyers. Following the consent process, three consecutive questionnaires (day 0 ,30, 90) were sent to the subjects. The data analysis will be done by using R program. The statistically significance in this study was classified at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residences who are currently studying in the department of Anesthesia

Exclusion Criteria:

* Refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - Anesthesia residences who are currently studying in the department of Anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Pre-class Self-directed learning time | 1 month before class
  Time spent for studying by the student, themselves, prior the simulation class
Post-class Self-directed learning time | upto 3 months after class
  Time spent for studying by the student, themselves, after the simulation class

SECONDARY OUTCOMES:
Knowledge retention | upto 3 months after class
  The percentage of knowledge (in pediatric anesthesia topic) retain after class
Level of self-confidence to treat the real patient | upto 3 months after class
  Level of self-confidence to treat the real patient after class

CONTACTS AND LOCATIONS:
Locations (1):
- Ngamjit Pattaravit, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided